CLINICAL TRIAL: NCT04470791
Title: Cryotherapy as a Coadjuvant in the Management of Crotaline Snakebite With F(ab')2 Antivenom: A Randomized Pilot Study.
Brief Title: Cryotherapy as a Coadjuvant in Crotaline Snakebite Management With Antivenom.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Juarez de Mexico (Other Government)
Responsible Party: Principal Investigator, Mario Adan Moreno Eutimio, Principal Investigator, Hospital Juarez de Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HJM 0142/16-R; HJM 0142/16-R (Other: Hospital Juárez de México)
Record Dates: First submitted 2020-07-06; First posted 2020-07-14 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Snake Bites
MeSH Terms: conditions — Snake Bites

STUDY DESIGN:
Intervention Model Description: A randomized pilot study was performed that included patients of both genders and over 18 years old with a snakebite of envenomation grade II who were admitted to the Clinical Toxicology Service of the Hospital Juárez de México.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding of the participants and interventionists was impossible, but the data analyst was blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F(ab')2 antivenom plus local cryotherapy. (Experimental): Group A: patients with a Crotalus snakebite, and grade II envenomation received F(ab')2 antivenom therapy and application of local cryotherapy.
  Interventions: Biological: F(ab)2 antivenom therapy (antivipmyn®).; Procedure: Local cryotherapy.
- F(ab')2 antivenom. (Active Comparator): Group B: patients who received only F(ab')2 antivenom therapy.
  Interventions: Biological: F(ab)2 antivenom therapy (antivipmyn®).

INTERVENTIONS:
Biological: F(ab)2 antivenom therapy (antivipmyn®). — Antivipmyn is an equine origin antivenom produced by Institute Bioclon in Mexico (Silanes Laboratories, México). The snake venoms used to create the F(ab')2 fragments are from Crotalus durissus and Bothrops asper. The number of doses of each patient depended on the classification and evolution, as indicated by the manufacturer for grade II envenoming: from 6 to 10 bottles of F(ab)2 antivenom therapy, intravenously, as an initial dose. One dose (bottle) consisted of 10 mL of polyvalent concentrated and modified horse antibodies treated by enzymatic digestion to neutralize the Bothrops asper venom to not less than 780 lethal dose 50 (LD50), and the Crotalus basiliscus venom to not less than 790 LD50.
Procedure: Local cryotherapy. — Interval cryotherapy consisted of applying a plastic bag (the size of the bag depending on the size of the lesion, approximately 28 x 46 cm) two-thirds filled with crushed ice (frapped) wrapped in a towel applied for 20 minutes every 4 hours at the site of the snakebite throughout the hospital stay. New ice bags were used after 4 hours.
  Arms: F(ab')2 antivenom plus local cryotherapy.

SUMMARY:
The study aimed to determine the effect of local cryotherapy as a coadjuvant in patients with snakebite treated with F(ab')2 therapy venom at the Hospital Juárez de Mexico.

DETAILED DESCRIPTION:
Introduction: Local cryotherapy induces vasoconstriction, which leads to a reduction in the inflammatory process. However, the efficacy of local cryotherapy as a coadjuvant in snakebite treatment with F(ab')2 antivenom is unknown.

Objective: Determine the effect of local cryotherapy as a coadjuvant in patients with snakebite treated with F(ab')2 therapy venom.

Material and methods: Subjects with snakebite envenomation accident grade II, according to the Christopher-Rodning classification, were enrolled from the Clinical Toxicology Service of the Hospital Juárez de México. One group of patients received F(ab')2 antivenom therapy (antivipmyn®) plus local cryotherapy, and another group received only F(ab')2 antivenom therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders and any age with a snake bite of poison grade II who were admitted to the Clinical Toxicology Service of the Hospital Juárez de México.

Exclusion Criteria:

* Patients of both genders and any age with a snake bite of poison grade I, III or IV who were admitted to the Clinical Toxicology Service of the Hospital Juárez de México.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Distal circumference of the affected limb on hospital admission. | Baseline.
  The circumference values of the injured limb were measured in the distal circumference (site farthest from the bite with the estimated maximum degree of edema, or at the end of the limb) on the affected extremity.
Proximal circumference of the affected limb on hospital admission. | Baseline.
  The circumference values of the injured limb were measured in the proximal circumference (5-10 cm from the site of the bite) on the affected extremity.
Middle circumference of the affected limb on hospital admission. | Baseline.
  The circumference values of the injured limb were measured in the middle circumference (intermediate measurement between the proximal and distal diameter) on the affected extremity.
Distal circumference of the affected limb on hospital admission. | up to 24 weeks
  The circumference values of the injured limb were measured in the distal circumference (site farthest from the bite with the estimated maximum degree of edema, or at the end of the limb) on the affected extremity. The measurement was recorded at the time of the patient's hospital discharge.
Proximal circumference of the affected limb on hospital admission. | up to 24 weeks.
  The circumference values of the injured limb were measured in the proximal circumference (5-10 cm from the site of the bite) on the affected extremity. The measurement was recorded at the time of the patient's hospital discharge.
Middle circumference of the affected limb on hospital admission. | up to 24 weeks.
  The circumference values of the injured limb were measured in the middle circumference (intermediate measurement between the proximal and distal diameter) on the affected extremity. The measurement was recorded at the time of the patient's hospital discharge.

SECONDARY OUTCOMES:
Hospital stay. | up to 24 weeks.
  The length of an inpatient episode of care, calculated from the day of admission to day of discharge, and based on the number of nights spent in hospital. Patients admitted and discharged on the same day have a length of stay of less than one day.

IPD SHARING:
Plan to Share IPD: No